CLINICAL TRIAL: NCT01445041
Title: Autologous Cord Blood Cells for Patients With HLHS: Phase I Study of Feasibility and Safety
Brief Title: Safety and Feasibility Study of Umbilical Cord Blood Cells for Infants With Hypoplastic Left Heart Syndrome
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Funding Period Ended
Sponsor: Michael Cotten (Other)
Responsible Party: Sponsor-Investigator, Michael Cotten, Associate Professor of Pediatrics, Duke University
Organization: Duke University (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00024650
Record Dates: First submitted 2011-09-15; First posted 2011-10-03 (Estimated); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Hypoplastic Left Heart Syndrome
Keywords: Hypoplastic Left Heart Syndrome; Autologous Umbilical Cord Blood; Newborn Infants
MeSH Terms: conditions — Hypoplastic Left Heart Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Single infusion of UCB (Experimental): (autologous red blood cell and volume reduced cord blood cells)
  Interventions: Biological: Autologous Umbilical Cord Blood
- Three infusions of UCB (Experimental): (autologous red blood cell and volume reduced cord blood cells)
  Interventions: Biological: Autologous Umbilical Cord Blood

INTERVENTIONS:
Biological: Autologous Umbilical Cord Blood — Infants who meet study enrollment criteria for hypoplastic left heart syndrome in the neonatal period will receive 1 infusion of their own volume reduced cord blood cells. The dose for each infusion is 5x10e7 cells/kg.
  Arms: Single infusion of UCB
Biological: Autologous Umbilical Cord Blood — Infants who meet study enrollment criteria for hypoplastic left heart syndrome in the neonatal period will receive 3 infusions of their own volume reduced cord blood cells. The first infusion will be a fresh, volume-reduced infusion and the subsequent infusions will be thawed and washed infusions. The dose for each infusion is 5x10e7 cells/kg.
  Arms: Three infusions of UCB

SUMMARY:
Further study details as provided by Duke University:

Purpose: To evaluate the feasibility and safety of collecting and infusing autologous umbilical cord blood (UCB) in newborn infants with hypoplastic left heart syndrome (HLHS).

Study Rationale and Hypotheses: The major goal of this study is to determine whether infusion of autologous UCB cells in neonates with hypoplastic left heart syndrome is feasible and safe. The rationale for the study and for the potential benefit of UCB is based upon the following hypotheses:

1. Infants with HLHS have significant neural injury evidenced from both prenatal and early antenatal brain MRI findings and infusion of UCB cells may lessen neural injury. Although the exact mechanism is unknown, UCB cell infusion may ameliorate neural injury via paracrine and anti-inflammatory effects that enhance post injury repair and may promote endogenous functional compensation of other cortical areas resulting in significant clinical improvements.
2. UCB cells may also enhance cardiac function, minimize scar formation, and reverse detrimental remodeling after cardiac injury.

DETAILED DESCRIPTION:
The purpose of this pilot study is to evaluate the safety and feasibility of infusions of autologous (the patient's own)umbilical cord blood cells in neonates with hypoplastic left heart syndrome. This is a prospective, randomized Phase I trial designed to assess the safety and feasibility of autologous UCB reinfusion in neonates with Hypoplastic Left Heart Syndrome (HLHS). Neonates who are identified prenatally as having a cardiac lesion consistent with HLHS will be referred to Duke Cardiology for further evaluation. If they meet inclusion criteria, UCB will be collected at the time of delivery and processed (red blood cell- and volume-reduced) for reinfusion. All enrolled infants will receive a dose of fresh UCB cells pre-operatively and ½ of the enrolled infants will be randomly selected to receive a second dose of frozen and thawed UCB cells after stage 1 palliation (5-35 days post-operatively) and a third dose of frozen and thawed UCB cells 2 to 4 weeks after the 2nd infusion. Neurodevelopmental outcome measures will be assessed at 1 month after discharge, at 4-6 months old and 12 months. The results of MRI's and echocardiograms that are obtained per clinical routine will be analyzed and described in study reports.

ELIGIBILITY:
Inclusion Criteria:

* Infants > 35 weeks gestational age.
* Diagnosis: Hypoplastic Left Heart Syndrome.
* Autologous umbilical cord blood available with a minimum total nucleated cell dose of 1 x 10e7 cells/kg.
* Parental Consent.

Exclusion Criteria:

* Chromosomal anomalies identified before the time of infusion.
* Chromosomal anomalies or congenital anomalies that would prohibit clinicians from initiating surgical repair of the congenital heart defect.
* Infant is determined by clinical staff to be non-viable and will not receive aggressive care. (No member on the study team will be involved in determining the viability of the neonate.)
* Autologous umbilical cord blood unit has any of the following:

  * Total nuclear cell count < 1 x 10e7.
  * Positive maternal infectious serology (except CMV).
  * Evidence of infectious contamination of the cord blood unit.
  * Evidence of genetic disease.
* Unable to obtain parental consent.
* Mother < 18 years old.

Max Age: 2 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 7 (Actual)
Dates: Start 2011-09-01 (Actual); Primary Completion 2016-04-15 (Actual); Study Completion 2016-04-15 (Actual)

PRIMARY OUTCOMES:
Adverse event rates occurring in the pilot study population. The investigators will compare infusion outcomes of infants infused with frozen cells and infants infused with non-frozen cells. | During Infusions (First 2 months of life)

SECONDARY OUTCOMES:
Feasibility and preliminary efficacy | 1 year
  Feasibility: volume of cord blood, cell viability, time to prepare/infuse fresh cells and frozen-thawed cells.
  Preliminary efficacy: neurodevelopmental outcomes at 9 - 12 months, cardiac function as assessed clinically.

CONTACTS AND LOCATIONS:
Overall Officials: Charles M Cotten, MD MHS, Principal Investigator — Duke University
Locations (1):
- Duke University, Durham, North Carolina, United States

REFERENCES:
- [Background] Martin PL, Carter SL, Kernan NA, Sahdev I, Wall D, Pietryga D, Wagner JE, Kurtzberg J. Results of the cord blood transplantation study (COBLT): outcomes of unrelated donor umbilical cord blood transplantation in pediatric patients with lysosomal and peroxisomal storage diseases. Biol Blood Marrow Transplant. 2006 Feb;12(2):184-94. doi: 10.1016/j.bbmt.2005.09.016. PMID 16443516
- [Background] Kurtzberg J, Lyerly AD, Sugarman J. Untying the Gordian knot: policies, practices, and ethical issues related to banking of umbilical cord blood. J Clin Invest. 2005 Oct;115(10):2592-7. doi: 10.1172/JCI26690. PMID 16200191
- [Background] Escolar ML, Poe MD, Provenzale JM, Richards KC, Allison J, Wood S, Wenger DA, Pietryga D, Wall D, Champagne M, Morse R, Krivit W, Kurtzberg J. Transplantation of umbilical-cord blood in babies with infantile Krabbe's disease. N Engl J Med. 2005 May 19;352(20):2069-81. doi: 10.1056/NEJMoa042604. PMID 15901860
- [Background] Staba SL, Escolar ML, Poe M, Kim Y, Martin PL, Szabolcs P, Allison-Thacker J, Wood S, Wenger DA, Rubinstein P, Hopwood JJ, Krivit W, Kurtzberg J. Cord-blood transplants from unrelated donors in patients with Hurler's syndrome. N Engl J Med. 2004 May 6;350(19):1960-9. doi: 10.1056/NEJMoa032613. PMID 15128896
- [Background] McGraw P, Liang L, Escolar M, Mukundan S, Kurtzberg J, Provenzale JM. Krabbe disease treated with hematopoietic stem cell transplantation: serial assessment of anisotropy measurements--initial experience. Radiology. 2005 Jul;236(1):221-30. doi: 10.1148/radiol.2353040716. PMID 15987975
- [Background] Mahle WT, Tavani F, Zimmerman RA, Nicolson SC, Galli KK, Gaynor JW, Clancy RR, Montenegro LM, Spray TL, Chiavacci RM, Wernovsky G, Kurth CD. An MRI study of neurological injury before and after congenital heart surgery. Circulation. 2002 Sep 24;106(12 Suppl 1):I109-14. PMID 12354718
- See also: Carolinas Cord Blood Bank web page — https://sites.duke.edu/ccbb/